CLINICAL TRIAL: NCT00204061
Title: Early Pharmacological and Psychological Intervention for Late Prodromal States of Psychosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); German Research Network On Schizophrenia (Network); Sanofi-Synthelabo (Industry); Department of Psychiatry University of Bonn (Other); Heinrich-Heine University, Duesseldorf (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Stephan Ruhrmann, Deputy Head of the Department of Psychiatry, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01 GI 9935 - P 1.1.3
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Schizophrenia; Psychoses
Keywords: schizophrenia; psychosis; ultra high risk; prodromal state; early intervention; amisulpride
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Prodromal Symptoms | interventions — Amisulpride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- supportive management (Placebo Comparator): needs-focused, unspecific supportive management
  Interventions: Behavioral: Supportive management
- amisulpride (Experimental): 24 months amisulpride 50 to 800 mg, needs-focused, unspecific supportive management.
  Interventions: Drug: Amisulpride

INTERVENTIONS:
Behavioral: Supportive management — The needs-focused intervention could include psychoeducation, crisis intervention, family counselling and assistance with education or work-related difficulties, according to need. Regular psychotherapy was not permitted.
  Other Names: Clinical Management
  Arms: supportive management
Drug: Amisulpride — Daily doses could range from 50 to 800 mg, with increments of 50 mg at first step and 100 mg at further steps. As a guideline, it was suggested that the dosage be increased as long as attenuated or brief limited intermittent positive symptoms were present. The interval between such steps should be at least 14 days if brief limited symptoms were absent and the APS score had improved.
  Other Names: Solian
  Arms: amisulpride

SUMMARY:
The study will provide an empirical basis for a pharmacological treatment option. An open-label, randomized, multi-centre parallel group design is used. An intensified clinical management (CM), which allows needs-based psychological crisis intervention, is compared to a combination of such a CM and the atypical neuroleptic amisulpride. The central hypothesis is that the combination of a clinical management with an atypical neuroleptic is the superior treatment.

DETAILED DESCRIPTION:
The first diagnosis of schizophrenia is preceded by a long lasting period comprising an untreated psychotic and a prodromal state. The duration of untreated psychosis correlates with a significant worsening of several outcome variables and persons fulfilling criteria of a prodromal state are already suffering from prodromal symptoms and from a significant deterioration of social and vocational functioning. However, a sufficient strategy for early intervention is still lacking. The study will provide an empirical basis for a pharmacological treatment option. An open-label, randomized, multi-centre parallel group design is used. An intensified clinical management (CM), which allows needs-based psychological crisis intervention, is compared to a combination of such a CM and the atypical neuroleptic amisulpride. For analysis 130 patients will be recruited within three years, the treatment period is two years.

ELIGIBILITY:
Inclusion Criteria:

1. General criteria

   * Age between 14 and 36 years
   * male or female, in- or outpatients
   * written informed consent, for patients below 18 years also signed by parents
2. Special criteria (present within the last three months prior to the study)

   * Attenuated Positive Symptoms (APS)
   * Presence of at least one of the following symptoms: ideas of reference, odd beliefs or magical thinking, unusual perceptual experiences, odd thinking and speech, suspiciousness or paranoid ideation
   * Symptoms have to appear several times per week for a period of at least one week

AND / OR

* Brief Limited Intermittent Psychotic Symptoms (BLIPS)
* Duration of episode less than one week, interval between episodes at least one week
* Symptoms resolve spontaneously
* Presence of at least one of the following symptoms: Hallucinations, Delusions, Formal thought disorder, Gross disorganized or catatonic behavior

Exclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders (DSM) IV diagnosis of schizophrenia, schizophreniform,schizoaffective, delusional or bipolar disorder, at any time of life.
* DSM-IV diagnosis of brief psychotic episode with a duration of more than one week, at any time time of life, or BLIPS within one week before inclusion.
* DSM-IV diagnosis of delirium, dementia, amnestic and other cognitive disorders, mental retardation, mental disorders due to a general medical condition or mental disturbances due to psychotropic substances.
* Abuse of alcohol or drugs within the last three months prior to the study; exception: cannabis user have to be drug-free during four weeks prior to the study. In case of drug abuse, it has to be determined, whether present prodromal symptoms appeared before any drug abuse; If not, symptoms have to be still present after a drug-free period of 3 months (hallucinogens, amphetamines), or four weeks (cannabis).

Ages: 14 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2001-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
improvement of risk related symptoms | 3, 6, 12, 24 months
  Decrease of symptom scores; complete remission of risk related symptoms

SECONDARY OUTCOMES:
Global functioning | 3, 6, 12, 24 months
  Increase of Global Assessment of Functioning (GAF) scores

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Klosterkötter, Professor, Study Chair — Department of Psychiatry and Psycotherapy University of Cologne
Locations (1):
- Department of Psychiatry and Psycotherapy University of Cologne, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- See also: Click here for more information about this study: Early pharmacological and psychological intervention for late prodromal states of psychosis — http://www.kompetenznetz-schizophrenie.de
- See also: Homepage of co-ordinating center — http://www.fetz.de